CLINICAL TRIAL: NCT03218306
Title: Surgical Pleth Index Guided Intraoperative Analgesia Versus Standard Clinical Approach During Desflurane Based General Anesthesia for Thyroidectomy
Brief Title: Surgical Pleth Index (SPI) Versus Standard Clinical Approach Analgesia
Acronym: SPIDER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Prof. Gabriele Finco, Professor of Anesthesiology and Intensive Care, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPI_3417
Record Dates: First submitted 2017-07-09; First posted 2017-07-14 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia; Pain; Surgery
Keywords: SPI; Remifentanil; Target controlled infusion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPI guided analgesia (Experimental): SPI ≤ 10 percentual points over the post-induction/pre-surgical incision value
  Interventions: Device: Surgical Pleth Index
- Clinical Guided Analgesia (Active Comparator): No SPI guidance
  Interventions: Other: Clinical guidance

INTERVENTIONS:
Device: Surgical Pleth Index — Effector site concentration of remifentanil based on SPI
  Arms: SPI guided analgesia
Other: Clinical guidance — Effector site concentration of remifentanil based on hemodynamic data
  Arms: Clinical Guided Analgesia

SUMMARY:
The study is aimed at confronting a surgical pleth index based protocol for intraoperative analgesia in a desflurane based general anesthesia for thyroidectomy, versus a standard clinical approach. A reduction in analgesic consumption and improvement in hemodynamics are expected.

ELIGIBILITY:
Inclusion Criteria:

* 18<age<80 years
* American society of anesthesiology (ASA) physical status I -II
* 6 hrs fasting

Exclusion Criteria:

* Arrhythmia or Pacemaker
* Central or peripheral nervous system or muscular disease
* Drugs active on autonomous nervous system (eg clonidine)
* Obesity (BMI >35)
* Chronic Pain
* Addictions or central nervous acting drugs use
* Hypertension (if not treated)
* Connective tissue disease
* Pregnancy
* Allergy or hypersensitivity to study drugs
* QT prolongation
* Absence of inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption | Intraoperative
  Cumulative remifentanil consumption throughout surgery

SECONDARY OUTCOMES:
Hemodynamics | intraoperative
  Cumulative number of episodes of hypotension or hypertension or brady/tachycardia
Desflurane | intraoperative
  Cumulative consumption of desflurane (ml) as measured by datex ohmeda aysis ventilator
Extubation delay | intraoperative
  Timespan between end of surgery and extubation
Post-operative analgesia 1 | 24 hr post operative
  Evaluate the total consumption of analgesics in the first 24 hours after surgery
Post-operative analgesia 2 | 24 hr post operative
  measure pain in the first post-operative day
Adverse reactions | 24 hr post operative
  Nausea and vomiting in the 1st post-operative day
Patient satisfaction | 24 hr post operative
  Evaluate on a 0-4 numeric scale patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Finco, MD, Study Director — University of Cagliari
Locations (1):
- Policlinico Duilio Casula, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided